CLINICAL TRIAL: NCT00831545
Title: Multicenter Phase 2 Evaluation of Temozolomide for Treatment of Brain Metastases of Either Malignant Melanoma, Breast and Non-small Cell Lung Cancer.
Brief Title: Study to Evaluate the Efficacy and Safety of Temozolomide in Subjects With Brain Metastases of Either Malignant Melanoma, Breast, or Non-small Cell Lung Cancer (P02064)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P02064
Record Dates: First submitted 2009-01-15; First posted 2009-01-29 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Metastases of Central Nervous System; Melanoma; Breast Neoplasm; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Melanoma; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Subjects with melanoma (Experimental)
  Interventions: Drug: Temozolomide
- Subjects with breast cancer (Experimental)
  Interventions: Drug: Temozolomide
- Subjects with non-small cell lung cancer (Experimental)
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — 150 mg/m2 given once a day for 7 consecutive days (Days 1 through 7) repeated every other week until disease progression or toxicity or for a maximum of one year. After amendment, schedule was modified: a second rest week was added after the second wash-out week (Days 1 through 7, 15 through 21 every 35).
  Other Names: SCH 52365

SUMMARY:
The study implies a 2 step study design. Patients are enrolled into 3 separate groups for melanoma, breast, and non-small cell lung cancer. In the first step, 21 patients per disease group are enrolled. If >=2 objective responses (SD, PR, or CR) out of 21 evaluable patients are observed, enrollment continues for other 45 patients as a whole, where response will be positively evaluated if >=10 patients will respond. If <2 objective responses out of 21 evaluable patients per disease group are observed, this(ese) group(s) will no longer be treated with temozolomide.

ELIGIBILITY:
Inclusion Criteria:

* Cytological/histological diagnosis of either melanoma, non-small cell lung cancer and breast;
* Brain metastases >=1 cm presenting or in progression following >=4 weeks time interval free from previous malignancy-specific chemotherapy, hormone therapy, or other medical therapies;
* Magnetic resonance imaging suspected brain metastases; patients with brain lesion(s) not univocal as brain metastases must have negative radiolabeled leukocyte brain scan to rule out infectious non-malignant disease; all neuroradiological studies (baseline and treatment outcome evaluation), except for emergency exams must be performed after 10 days of unchanged schedule of dexamethasone, and obtained in the axial-coronal-sagittal planes in T1 and T2 before and after gadolinium enhancement.
* Presence of al least one bidimensionally measurable and not previously irradiated metastasis.
* Age <=70 years.
* Performance status 0-2 (ECOG-WHO scale).
* Blood leukocytes >=3.5 x 10^9/L and platelets >=100 x 10^9/L.
* Bilirubin <=25 M/L.
* Seric transaminases <=2 x upper limit of normal values.
* Creatinine <=150 M/L, creatinine clearance >=60 mL/min.
* Signed written informed consent.

Exclusion Criteria:

* Diabetes not allowing administration of adequate doses of dexamethasone at least during the first 2 months of treatment.
* Previous whole brain irradiation.
* Brain metastases eligible to neurosurgery or stereotactic radiation therapy.
* Previous or current malignancies at other sites with the exception of adequately treated in situ carcinoma of the cervix or basal and squamous carcinoma of the skin.
* Pregnant or nursing women.
* Acute infection requiring intravenous antibiotics.
* Severe vomiting or medical condition which could interfere with oral medication intake.
* Anticonvulsant chronic therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2000-12-01 (Actual); Primary Completion 2006-10-20 (Actual); Study Completion 2006-10-20 (Actual)

PRIMARY OUTCOMES:
Best response related to brain metastases observed during the study period. | After 2 months of initial treatment. If response or stable disease evaluations were performed every 3 months. Subsequently, an additional check up was added by amendment: a follow up check was performed after 4 weeks.

SECONDARY OUTCOMES:
Progression-free survival, brain progression-free survival, and overall survival. | After 2 months of initial treatment. If response or stable disease evaluations were performed every 3 months. Subsequently, an additional check up was added by amendment: a follow up check was performed after 4 weeks.
Adverse events according to NCI CTC grading system of toxicity. | Throughout the study.

REFERENCES:
- [Result] Siena S, Crino L, Danova M, Del Prete S, Cascinu S, Salvagni S, Schiavetto I, Vitali M, Bajetta E. Dose-dense temozolomide regimen for the treatment of brain metastases from melanoma, breast cancer, or lung cancer not amenable to surgery or radiosurgery: a multicenter phase II study. Ann Oncol. 2010 Mar;21(3):655-661. doi: 10.1093/annonc/mdp343. Epub 2009 Sep 18. PMID 19767314
- Available data/document: CSR Synopsis Links — http://www.merck.com/clinical-trials/policies-perspectives.html